CLINICAL TRIAL: NCT06307873
Title: Comparison of the Effects of Sacrospinous Fixation and V-notes Lateral Suspension Operations on Anatomical Recovery, Effectiveness and Quality of Life.
Brief Title: Comparison of the Effects of Sacrospinous Fixation and V-notes Lateral Suspension Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREH.
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-12

CONDITIONS: Genital Prolapse, Unspecified
Keywords: sacrospinous fixation; v-notes lateral suspension; genital prolapse
MeSH Terms: interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients undergone Sacrospinous Fixation operation (Active Comparator)
  Interventions: Diagnostic Test: pre and post operative POP-Q results; Behavioral: pre and post operative PİSQ-12 results
- patients undergone V-notes Lateral Suspension Operation (Active Comparator)
  Interventions: Diagnostic Test: pre and post operative POP-Q results; Behavioral: pre and post operative PİSQ-12 results

INTERVENTIONS:
Diagnostic Test: pre and post operative POP-Q results — Comparison of pre and postoperative POP-Q values of the patients undergone Sacrospinous Fixation operation and V-notes Lateral Suspension Operation
Behavioral: pre and post operative PİSQ-12 results — Comparison of pre and postoperative PİSQ-12 values of the patients undergone Sacrospinous Fixation operation and V-notes Lateral Suspension Operation

SUMMARY:
Comparison of the effects of sacrospinous fixation and v-notes lateral suspension operations on anatomical recovery, effectiveness and quality of life in a training and research hospital gynecology and obstetrics clinic.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 35-75 patients without pelvic mess, servical or endometrial lesion

Exclusion Criteria:

* patients with pelvic mess, servical or endometrial lesion patient with diagnosed endometrial cancer

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Pre and post operative assessment of POP-Q measurements | 1 year
  POP-Q values of patients before and after Sacrospinous Fixation and V-notes Lateral Suspension Operations on Pelvic Organ Prolapse will be compared
Pre and post operative assessment of Pelvic Organ Prolapse / Incontinence Sexual | 1 year
  PISQ-12 values of patients before and after Sacrospinous Fixation and V-notes Lateral Suspension Operations on Pelvic Organ Prolapse will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)